CLINICAL TRIAL: NCT02055729
Title: Changes in Cutaneous, Digestive and Urinary Bacterial Flora Among Patients With Pelvic Bedsores: a Prospective Pilot Study
Brief Title: Changes in Bacterial Flora Among Patients With Pelvic Bedsores: a Prospective Pilot Study
Acronym: EscaFlor
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: PERSE (Prévention, Education, Recherche, Soins, Escarres) Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/CDR-01; 2014-A00534-43 (Other: RCB number)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Bedsore
Keywords: bedsore; bacteria; colonization; ecology
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bedsore superficial (swabbing) and deep (punch biopsies) samples are retained; stool and urine samples are retained. DNA extraction is aimed at describing microbial communities.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The proposed study is a prospective, single-center pilot study lasting 28 days. Our goal is to study the temporal evolution of the bacterial communities present in the skin and digestive flora (stool) of spinal cord injured persons having one or more sacral bedsores. The study timespan can include treatment initiation, notably of antibiotics. Urinalysis for studying urinary flora will simultaneously occur.
  For a description of the study population, see the inclusion/exclusion criteria.
  Intervention: Superficial bedsore sample Intervention: 3mm tissue punch biopsy Intervention: Stool sample Intervention: Urine sample
  Interventions: Biological: 3mm tissue punch biopsy; Biological: Superficial bedsore sample; Biological: Stool sample; Biological: Urine sample

INTERVENTIONS:
Biological: 3mm tissue punch biopsy — Bacterial samples will be collected using deep level tissue biopsy using a Steifel punch of 3 mm in diameter (days 0 and 28).
Biological: Superficial bedsore sample — Bacterial samples will be taken from the surface of the bedsore via swabbing. (days 0 & 28)
Biological: Stool sample — Stool samples will be collected on days 0 and 28.
Biological: Urine sample — Urine samples will be collected on days 0 and 28.

SUMMARY:
The main objective of this study is to characterize the evolution (over a period of 28 days) of superficial and deep bacterial skin flora in patients with stage 3 or 4 sacral pressure ulcers (bedsores). Changes in terms of pathogenic, potentially pathogenic and non-pathogenic bacterial species at the intra-individual and population levels.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To compare bacterial communities collected from superficial versus deep samples of stage 3 or 4 sacral bedsores using metagenomics and standard culturing methods.

B. To characterize the evolution of digestive bacterial flora in the same patients over a period of 28 days. Changes in terms of pathogenic, potentially pathogenic and non-pathogenic will be described, as well as the appearance of resistance phenotypes.

C. To characterize the evolution of urinary bacterial flora in the same patients over a period of 28 days. Changes in terms of pathogenic, potentially pathogenic and non-pathogenic will be described, as well as the appearance of resistance phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* The patient was correctly informed about study implementation, its objectives, constraints and patient rights
* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 28 days of follow-up
* The patient has one or more pelvic pressure ulcers (bedsores)(stage 3 or 4 only). Note: Patients with bedsores of varying stage will be included for the wound corresponding to the highest stage. If the patient has multiple bedsores of the same stage, the deepest wound will be selected.
* The patient requires a modern wound dressings (i.e. not tulle or gauze) without added bactericidal or antibiotic elements
* The patient is hospitalized ant the Propara neurological rehabilitation center (Montpellier, France)
* The patient has not received antibiotics in the last 14 days.

Exclusion Criteria:

* The patient is participating in another study, or has participated in another study in the last 3 months
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient is already included in the present study
* The patient has sacral pressure ulcers of only stages 1 or 2, or does not have a sacral pressure ulcer
* Patient under curative anticoagulation
* Patient who received antibiotics within 14 days before inclusion (however, after inclusion, the patient can be treated with antibiotics if necessary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients hospitalized in the Propara neurological rehabilitation (Montpellier, France) having at least one stage 3 or 4 bedsore in the pelvic region.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
List of pathogenic, potentially pathogenic and commensal bacterial species in superficial and deep bedsore samples | Baseline (day 0)
  At the individual level
List of pathogenic, potentially pathogenic and commensal bacterial species in superficial and deep bedsore samples | Day 28
  At the individual level
Percentage of pathogenic, potentially pathogenic, and commensal bacterial species in superficial and deep bedsore samples | baseline (day 0)
  Calculated over the entire study population
Percentage of pathogenic, potentially pathogenic, and commensal bacterial species in superficial and deep bedsore samples | Day 28
  Calculated over the entire study population

SECONDARY OUTCOMES:
Classification of bacteria present according to respiratory type, gram negative/positive, shape, and resistance phenotypes. | baseline (Day 0)
  Based on superficial and deep bedsore samples.
Classification of bacteria present according to respiratory type, gram negative/positive, shape, and resistance phenotypes. | Day 28
  Based on superficial and deep bedsore samples.
List of pathogenic, potentially pathogenic and commensal bacterial species in stool samples | baseline (day 0)
List of pathogenic, potentially pathogenic and commensal bacterial species in stool samples | Day 28
List of pathogenic, potentially pathogenic and commensal bacterial species in urine samples | baseline (day 0)
List of pathogenic, potentially pathogenic and commensal bacterial species in urine samples | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Dunyach-Remy, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (4):
- France (4):
  - Centre Mutualiste Neurologique Propara, Montpellier
  - Laboratoire d'Etude et de Recherche en Environnement et Santé, Unité Biodiagnostic, UNIMES, Nîmes
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Unité U1047 "Bacterial virulence and infectious diseases", UFR de Médecine, Nîmes

REFERENCES:
- [Derived] Fayolle M, Morsli M, Gelis A, Chateauraynaud M, Yahiaoui-Martinez A, Sotto A, Lavigne JP, Dunyach-Remy C. The Persistence of Staphylococcus aureus in Pressure Ulcers: A Colonising Role. Genes (Basel). 2021 Nov 25;12(12):1883. doi: 10.3390/genes12121883. PMID 34946833